CLINICAL TRIAL: NCT07345598
Title: Training in Central Venous Catheter Care: Effects on Knowledge and Infection Prevention Behaviors of Pediatric Oncology Nurses
Brief Title: Central Venous Catheter Care Training for Pediatric Oncology Nurses
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Collaborators: Acibadem Maslak Hospital (Other)
Responsible Party: Principal Investigator, Emine I Yıldız, Principal Investigator, Nurse, Fenerbahce University, Fenerbahce University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FBU-YILDIZ-001
Record Dates: First submitted 2025-09-12; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Cancer; Pediatric Oncology; Central Venous Catheter; Central Venous Catheter Placement; Central Venous Catheter Exit Site Infection
Keywords: Pediatric Nursing; Central venous catheter placement; Central Venous Catheter Exit Site Infection; Nurse training; hand hygiene; knowledge; infection prevention; clinical education; quasi-experimental study
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: All participants will receive central venous catheter care training follewed by evaluation of knowledge and infection prevention behaviors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training Group (Experimental): Participants in this arm will receive the central venous catheter care training program, including theoretical education, video demonstration, and hansd-on practice.
  Interventions: Other: CVC Care Training

INTERVENTIONS:
Other: CVC Care Training — The intervention consists of an educational training program including a PowerPoint presentation, training video, and hands-on practice with a mannequin. Data collection tools include the Sociodemographic Information Form, the Evidence-Based Guidelines Knowledge Test, and the Nurses' Observation Questionnaire on Infection Control and Prevention.

SUMMARY:
The knowledge level of nurses regarding care techniques plays a crucial role in the prevention of central venous catheter-related infections. This study was designed to evaluate the effect of training on central venous catheter care (CVCC), provided to nurses caring for pediatric oncology patients, on their knowledge level and infection prevention behaviors. The study aims to determine the effectiveness of an educational program intended to enhance nurses' knowledge and practical skills in preventing CVC-related infections, thereby contributing to evidence-based practices that improve patient safety.

DETAILED DESCRIPTION:
Quasi-experimental, pre-test/post-test desing with a control group. Central catheters are frequently used in hematology and oncology clinics. They are invasive devices employed in hospitalized patients for fluid therapy, drug administration, blood transfusions, total parenteral nutrition, and hemodynamic monitoring. In addition to enabling the effective continuation of treatment, they provide patients with a more comfortable therapeutic experience.

Proper maintenance of catheters is crucial for treatment continuity. Despite their medical advantages, central venous catheters (CVCs) are associated with complications such as infection, hemorrhage, and thrombosis. When central venous catheterization and catheter care are performed by inexperienced personnel or teams, the risk of catheter colonization and infection increases. Furthermore, if the catheter remains in place for more than five days, the risk of infection is eight times higher in groups using gauze dressings and microporous tape.

CVC-related infection is a significant cause of morbidity and mortality in immunocompromised children and adults, with infection-related mortality estimated between 12% and 25%. Recent studies have demonstrated that standardization of aseptic techniques and the provision of regular training reduce the risk of infection, while catheter insertion and maintenance by inexperienced personnel increase the likelihood of colonization or infection.

Nurses are key personnel both during central venous catheter insertion and in ensuring catheter care is maintained with aseptic technique . Regular training of healthcare professionals responsible for catheter insertion and care, ensuring compliance with hand hygiene, and adopting maximum barrier precautions during insertion (use of sterile gloves, gown, sterile drape covering the insertion site, mask, and cap) are recommended. In addition, the use of >0.5% chlorhexidine-alcohol combinations for skin antisepsis, routine use of chlorhexidine/antiseptic-impregnated catheters, and chlorhexidine-impregnated dressings are advised.

There are various nursing care practices aimed at preventing CVC-associated infections. It has been recommended that healthcare professionals conduct high-level evidence clinical studies to evaluate the effectiveness of these practices on infection, develop clinical protocols that may serve as guidelines for CVC care, and monitor these protocols regularly. Many healthcare institutions provide not only initial training for newly employed staff but also refresher training for existing personnel. Since aseptic techniques are complex, nurses need to complement their education with practical training to strengthen their knowledge and skills. CVC-associated infections remain an important risk factor; however, with properly planned training, nurses' knowledge of current guidelines and their compliance with them should be periodically evaluated . Educational programs provided to nurses should be didactic, evidence-based, and structured with appropriate content and timing.

Nursing is an applied profession that requires meaningful integration of theoretical knowledge and practical skills. Therefore, this study was designed to evaluate the effect of theoretical and practical training on central venous catheter care, provided to nurses caring for pediatric oncology patients, on their knowledge level and infection prevention behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Provided care to a pediatric oncology patient at least once
* Performed a procedure via a central venous catheter on a pediatric oncology patient
* Voluntarily signed the informed consent form

Exclusion Criteria:

* Not having previously performed a procedure via a central venous catheter

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-22 (Estimated); Primary Completion 2026-05-22 (Estimated); Study Completion 2026-06-22 (Estimated)

PRIMARY OUTCOMES:
Change in Infection Prevention Behaviors | During the 4 weeks before training (baseline) and during the 4 weeks after completion of the training program
  Measured by the Nurses' Observation Checklist for Infection Control and Prevention (19 items). Higher scores indicate better infection prevention practices. Nurses will be observed before and after the training.
Change in Knowledge Level of Nurses | At baseline (pre-training) and on the same day immediately after completion of the training
  Measured by the Evidence-Based Guidelines Knowledge Test (10 questions). Higher scores indicate greater knowledge. Nurses will complete the test before and after the training.

SECONDARY OUTCOMES:
Post-Training Observation of Infection Prevention Behaviors | At 4 weeks after completion of the training program
  Nurses will be observed in their clinical practice environment after completing the training program. Observations will be conducted by the principal investigator and an independent observer using the Nurses' Observation Checklist for Infection Control and Prevention (19 items). Higher scores indicate better infection prevention practices. Scores will be recorded as post-training results.

CONTACTS AND LOCATIONS:
Overall Officials: Yagmur Sancı, Assistant Professor, Study Director — Fenerbahce University
Locations (1):
- Acıbadem Maslak Hospital - Pediatric Oncology Unit, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be available from the corresponding author upon reasonable request for academic and scientific research purposes.
Supporting Information: Study Protocol
Time Frame: 6 months after publication-5 years
Access Criteria: De-identified IPD will be available to qualified researchers for academic and scientific purposes. Access will be granted upon reasonable request to the corresponding author, subject to approval of a research proposal and compliance with institutional ethical standards.

DOCUMENTS (1):
  • Study Protocol (2025-09-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT07345598/Prot_000.pdf